CLINICAL TRIAL: NCT02712190
Title: Evaluation of Prolonged Apnea Supported by High Frequency Non-invasive Ventilation.
Acronym: ANIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Adam Ogna, MD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ANIV
Record Dates: First submitted 2016-03-10; First posted 2016-03-18 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Non-invasive Ventilation; High-frequency Ventilation; Healthy Volunteer; Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low - High frequence sequence (Experimental): High-Frequency non-invasive ventilation (HF-NIV) with 2 different settings, sequence of respiratory rate 250/min and respiratory rate 500/min
  Interventions: Device: High-frequency non-invasive ventilation
- High - Low frequence sequence (Experimental): High-Frequency non-invasive ventilation (HF-NIV) with 2 different settings, sequence of respiratory rate 500/min and respiratory rate 250/min
  Interventions: Device: High-frequency non-invasive ventilation

INTERVENTIONS:
Device: High-frequency non-invasive ventilation — Comparison of 2 different settings of HF-NIV
  Other Names: HF-NIV

SUMMARY:
The purpose of the study is to assess the efficacy of high-frequency non-invasive ventilation on apnea duration, carbon dioxide clearance and oxygen delivery in healthy subjets and patients with lung disease.

DETAILED DESCRIPTION:
High frequency ventilation (HF-V) allows to ensure oxygen delivery and carbon dioxide clearance despite the absence of thoracic movement in anesthetized, invasively ventilated subjects. This same technique could be applied by a non-invasive interface (HF-NIV), allowing to obtain a prolonged apnea (absence of thoraco-abdominal respiratory movements) in awaken subjects. Such an application would be of interest for several clinical applications, e.g. lung imaging and radio-therapy treatment on lung cancer. The purpose of the study is to assess the effect of different HF-NIV setting on the apnea duration, carbon dioxide clearance and oxygen delivery in healthy subjets and patients with lung diseases.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjets : normal respiratory function and no known lung disease
* lung disease patients : chronic obstructive pulmonary disease, Sarcoidosis, Cystic fibrosis
* age >=18y

Exclusion Criteria:

* increased pneumothorax risk under positive pressure ventilation
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Duration of apnea | 1 study session (2 hours)
  Duration of apnea according to the different settings of the HF-NIV, defined as absence of thoraco-abdominal respiratory movements

SECONDARY OUTCOMES:
Transcutaneous carbon dioxide partial pressure | 1 study session (2 hours)
  Evolution of transcutaneous carbon dioxide partial pressure (TcCo2)
Oxygen saturation of arterial blood | 1 study session (2 hours)
  Evolution of oxygen saturation, measured by pulse-oximetry (SatO2)
Lung volume | 1 study session (2 hours)
  Evolution of lung volume
Subjective tolerance | 1 study session (2 hours)
  Subjective tolerance of the HF-NIV (questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Alban Lovis, Principal Investigator — Service de Pneumologie - CHUV
Locations (1):
- Service de Pneumologie - Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No